CLINICAL TRIAL: NCT07379372
Title: Bladder Overactivity and Post-Botulinum Toxin Telemonitoring: a Randomized, Controlled, Superiority Trial
Brief Title: Bladder Overactivity and Post-Botulinum Toxin Telemonitoring
Acronym: VESIC@HOME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 38RC24.0402
Record Dates: First submitted 2025-12-19; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Overactive Bladder
Keywords: urinary incontinence; botulinum toxin; connected urinary incontinence
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence | interventions — Home Care Services

STUDY DESIGN:
Intervention Model Description: prospective, randomized and controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hospital based follow-up (No Intervention): The patient must arrive with a full bladder (a minimum volume of 150 mL, including both the voided volume and the post-void residual), refrain from voiding until urinating into the uroflowmeter, have completed their bladder diary at home beforehand (measuring with a graduated container over 3 days and 3 nights), have filled out the EQ-5D-5L (quality of life), USP (urinary symptoms), and PGI (post-treatment global impression of improvement) questionnaires, and bring them along
- home based follow-up group (Experimental): A nurse from the provider will bring the equipment required for the different measurements (Homeflow®) and explain its use to the patient. The nurse will also give the patient the EQ-5D-5L (quality of life), USP (urinary symptoms), and PGI (post-treatment global impression of improvement) questionnaires in paper format. A first assessment of the PVR may already be performed. The nurse will return to collect the equipment and questionnaires and to perform a PVR measurement 72 hours later. The recorded data are transmitted directly to the physician, who can view them on their computer (a dedicated secure application provided with the Homeflow solution) and export them in PDF format to add them to the patient's file."
  Interventions: Other: home care

INTERVENTIONS:
Other: home care — 6-week follow-up visit: At home (The service provider will bring the necessary equipment for the various measurements and the questionnaires, and will explain their use to the patient. The provider will return to collect the equipment and perform a post-void residual (PVR) measurement 72 hours later.)
  Arms: home based follow-up group

SUMMARY:
Prospective, randomized, controlled, single-center study to compare the feasibility of home monitoring for patients receiving intradetrusor botulinum toxin injections with that of the usual hospital-based follow-up.

DETAILED DESCRIPTION:
Overactive bladder (OAB) affects seventeen percent of the French population and is characterized by a sudden urge to urinate, urinary frequency, with or without incontinence.

Botulinum toxin, injected into the bladder every 6 to 12 months, is an effective treatment. In 2022, more than 10,000 injections were performed in France (ATIH data). At the Grenoble University Hospital (CHUGA), 190 injections were recorded in 2018 and 300 in 2023. As elsewhere, the active patient cohort is increasing exponentially.

Treatment efficacy is assessed using a voiding diary (VD): a three-day record of each voiding episode with bladder capacity, frequency, and leakage. It is essential to detect the onset of voiding dysfunction through uroflowmetry and ultrasound measurement of post-void residual (PVR) at 6 weeks after injection (peak diffusion and efficacy). This allows determining the dose and frequency of reinjections. The goal is to improve quality of life, but also to protect the upper urinary tract, particularly in neurogenic bladders.

These 300 annual injections require 300 follow-up consultations, but many data points are often missing. Indeed, patients currently often attend post-injection consultations without a voiding diary and with a non-empty bladder… It is therefore important to improve this follow-up.

With our VESIC@HOME project, we aim to provide patients with the services of the home-care provider IC@dom and, thanks to suitable connected tools (Homeflow®), collect VD and uroflowmetry/PVR at home, as well as quality-of-life questionnaires, thereby improving data completeness under more physiological and comfortable conditions for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a neurogenic bladder or idiopathic overactive bladder.
* Patient treated with intradetrusor botulinum toxin injection as part of their usual care, whether performing spontaneous voiding or self-catheterization.
* Patient whose residence allows a home visit by a service provider within the area covered by the AGIR à dom group.
* Patient affiliated with the social security system.
* Patient willing to provide informed consent

Exclusion Criteria:

* Persons covered under Articles L1121-5 to L1121-8 of the French Public Health Code (CSP), corresponding to all protected persons: pregnant or postpartum women, breastfeeding mothers, individuals deprived of liberty by judicial or administrative decision, persons receiving psychiatric care under Articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of Article L. 1121-8, individuals admitted to a healthcare or social facility for purposes other than research, minors, persons under legal protection, or individuals unable to give consent.
* Staff members with a hierarchical relationship with the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2031-03-02 (Estimated)

PRIMARY OUTCOMES:
To compare the feasibility of home follow-up in patients receiving intradetrusor botulinum toxin injections with that of the usual hospital-based follow-up | at 8 weeks
  Rate of completeness of data collected at home compared with data collected in the hospital setting.
  To be considered complete, the data must include:
  The 3-day/3-night bladder diary (including the time and volume of each void); a diary is considered complete even if 3 measurements over the 72-hour period are missing (this accounts for possible patient appointments).
  The urinary symptom questionnaire (Urinary Symptom Profile, USP);
  Uroflowmetry and post-void residual measurements (only for patients who do not perform intermittent self-catheterization).
  All of these data are necessary to address the objective. We cannot separate them, as they serve the same objective.

SECONDARY OUTCOMES:
Compare urinary symptoms according to the type of follow-up. | at 8 weeks
  USP (urinary symptoms profil) questionnaire score at 6-8 weeks post-injection. Score ranging from 0 to 33; the higher the score, the more incontinent the patient is.
Compare functional outcomes ( Normal bladder emptying with not significant post-void residual) according to the type of follow-up in patients with spontaneous voiding. | at 8 weeks
  Uroflowmetry results and post-void residual (PVR) at 6-8 weeks post-injection both criteria are required to evaluate the same outcome
Compare complications according to the type of follow-up. | at 8 weeks
  Adverse events occurring up to 6-8 weeks post-injection: urinary retention requiring self- or caregiver catheterization, symptomatic urinary tract infection with or without fever.
Compare overall quality of life according to the type of follow-up. | at 8 weeks
  EQ-5D-5L scale at 6-8 weeks post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: caroline ct thuillier, physician, Principal Investigator — university grenoble hospital

IPD SHARING:
Plan to Share IPD: No